CLINICAL TRIAL: NCT05609279
Title: Metabolic Phenotypes and Heterogeneity in Disease Burden Risk in Type 1 Diabetes
Acronym: JDRF-COE
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, Rodica Pop-Busui, Professor of Internal Medicine, University of Michigan
Other Study IDs: HUM00185622
Record Dates: First submitted 2022-11-01; First posted 2022-11-08 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Diabetes Mellitus
Keywords: diabetes; type-1 diabetes mellitus; endocrinology
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Laboratory Measures:
  Blood and urine will be obtained for several laboratory tests including hemoglobin A1c (HbA1c), Lipid panel, Kidney Function. Urine will be obtained for urine microalbumin and protein measurements.
  Biosamples collection:
  Fasting blood and urine will also be collected for biomarkers assessments. With participant approval the study team will store sample for unspecified future research. This future research may involve DNA testing. Total blood storage at each in person visit will be 15mL. Total urine storage at each in person visit will be 50mL.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study focuses on individuals with type 1 diabetes (T1D) and seeks to comprehensively study and understand several aspects of T1D including: susceptibility to hypoglycemia (low blood sugar) and improvement in hypoglycemia risk using of advanced diabetes technologies, such as continuous glucose monitoring (CGM); the differences among individuals with T1D in the risk of chronic complications, and minimize the psychosocial impact of T1D.

DETAILED DESCRIPTION:
The study seeks to comprehensively study and understand several aspects of type 1 diabetes (T1D) including: the risk of low blood sugar and how that may be improved with new technologies; the variability (heterogeneity) among individuals in their risk of diabetes complications, and factors that could impact the psychosocial burdens of having T1D. The investigators want to learn of there are patient-specific systemic metabolomic profiles (substances detected in blood or urine) that lower the risk for hypoglycemia. Metabolomic analyses will be used to discover biological markers that could predict who is most likely to get diabetes complications, and how these risks might be changed, for example, by developing treatments targeted specifically to those biological markers. The investigators also plan to describe the relationship between metabolomic profiles, psychosocial states and cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* All participants with type 1 diabetes
* Previous enrollment and participation in the University of Michigan T1D cohorts (Natural History of Myocardial Dysfunction in T1D (HUM00036408); Targeting Inflammation with Salsalate in a T1D(HUM00169353); Preventing Early Renal Loss with Allopurinol in T1D (HUM00080944); and Tissue Specific Metabolic Reprogramming (HUM00060967)).
* Willing and able to participate in the study procedures described in the consent form.
* Willing to sign a written or electronic informed consent, including authorization to release health information.
* Fluent in spoken and written English.
* Willing to carry around their mobile phone/study mobile phone during the 14-day home monitoring period with daily access to cellular or WiFi connectivity.

Exclusion Criteria:

* Any social or medical condition that would, in the opinion of the Principal Investigator (PI), prevent complete participation in the study or would pose significant hazard to the subject's participation.
* Skin conditions or diseases that would interfere with the Continuous Glucose Monitor (CGM) sensor placement or accuracy (such as extensive psoriasis, extensive eczema, scarring, etc.)
* Scheduled X-ray, MRI, CT scan, or high-frequency electrical heat (diathermy) treatment during the period of CGM wear (or any other activity that would necessitate CGM sensor removal) that cannot be scheduled around or accommodated within the study assessment windows.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All participants with type 1 diabetes previously enrolled and that participated in the University of Michigan T1D cohorts
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-02-18 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Proportion of enrolled participants providing serum samples for metabolomic analysis | 3 years
  Metabolomic samples will be requested from all study participants at the first (Visit 1) and last (Visit 3) study visit. The last study visit will be within 3 years of the first.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided